CLINICAL TRIAL: NCT00883727
Title: A Randomized, Double Blind, Multicentric, Placebo Controlled, Single Dose, Phase - i/ii Study Assessing the Safety and Efficacy of Intravenous ex Vivo Cultured Adult Allogenic Mesenchymal Stem Cells in Patients With st Elevated Acute Myocardial Infarction (Stemi)
Brief Title: Ex Vivo Cultured Bone Marrow Derived Allogenic MSCs in AMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRPL/AMI/07-08/001
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Myocardial Infarction
Keywords: mesenchymal stem cells; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stem cells (Experimental)
  Interventions: Drug: Stem cell
- Placebo (Placebo Comparator)
  Interventions: Drug: Plasmalyte A

INTERVENTIONS:
Drug: Stem cell — IV infusion of stem cells
  Arms: stem cells
Drug: Plasmalyte A — IV infusion
  Arms: Placebo

SUMMARY:
This clinical trial aims to find out the safety and efficacy of adult mesenchymal stem cells in patients with myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI aged between 20 and 70 years, either males or females with non-child bearing potential, after 2 days of successful PCI.
* Patient has global left ventricular systolic dysfunction with an ejection fraction of <50% and >30%.
* ECG with sign of acute anterior MI with ST-elevation ≥ 2 mm in at least 2 of the following leads I, AVL, V1-V6, or ECG with sign of acute inferoposterior MI with ST-elevation ≥1 mm on all of the following leads- II, III, V5-V6 or STelevation ≥ 2 mm in at least 2 of the leads.
* The target lesion located in the proximal section of the left anterior descending, left circumflex or right coronary artery.
* Patient with acute myocardial infarction within 10 days prior to IP administration.
* Normal liver and renal function.
* Able to understand study information provided to him.
* Able to give voluntary written consent.

Exclusion Criteria:

* History of acute/chronic inflammatory condition or severe aortic stenosis or insufficiency; severe mitral stenosis or severe mitral insufficiency.
* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year.
* Advanced renal dysfunction and creatinine ≥ 2mg%.
* Advanced hepatic dysfunction.
* Have clinically serious and/or unstable intercurrent infection, medical illnesses or conditions that are uncontrolled or whose control, in the opinion of the Investigator, may be jeopardized by participation in this study or by the complications of this therapy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
AE and ECG parameters | 6 months

SECONDARY OUTCOMES:
Regional myocardial perfusion and infarct size | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sreenivas Kumar, MD, DM, Principal Investigator — Care Hospital, Hyderabad; Satya Gupta, Principal Investigator — SAL Hospital, Ahmedabad; R Keshava, MD, DM, Principal Investigator — Bhagwan Mahaveer JAin Hospital, Bangalore; Prakash VS, MD., DM, Principal Investigator — MS Ramaiah Memorial Hospital, Bangalore
Locations (4):
- India (4):
  - Care Hospital, Hyderabad, Andhra Pradesh
  - SAL Hospital and Medical Institute, Ahmedabad, Gujarat
  - MS Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Bhagawan Mahaveer Jain Heart Centre, Bangalore, Karnataka

REFERENCES:
- [Derived] Chullikana A, Majumdar AS, Gottipamula S, Krishnamurthy S, Kumar AS, Prakash VS, Gupta PK. Randomized, double-blind, phase I/II study of intravenous allogeneic mesenchymal stromal cells in acute myocardial infarction. Cytotherapy. 2015 Mar;17(3):250-61. doi: 10.1016/j.jcyt.2014.10.009. Epub 2014 Dec 4. PMID 25484310